CLINICAL TRIAL: NCT00148798
Title: Open, Randomized, Controlled, Multicenter Phase III Study Comparing Cisplatin/Vinorelbine Plus Cetuximab Versus Cisplatin/Vinorelbine as First-line Treatment for Patients With Epidermal Growth Factor Receptor Expressing (EGFR-expressing) Advanced NSCLC.
Brief Title: Study of Cisplatin/Vinorelbine +/- Cetuximab as First-line Treatment of Advanced Non Small Cell Lung Cancer (FLEX)
Acronym: FLEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 62202-046
Record Dates: First submitted 2005-09-07; First posted 2005-09-08 (Estimated); Results first posted 2011-10-04 (Estimated); Last update posted 2014-06-25 (Estimated); Status verified 2014-06

CONDITIONS: Non Small Cell Lung Cancer (NSCLC)
Keywords: Cetuximab; Non small cell lung cancer; Lung cancer; Cisplatin/vinorelbine; Monoclonal antibody; Erbitux
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Cetuximab; Cisplatin; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab plus chemotherapy (Experimental): cetuximab + cisplatin + vinorelbine
  Interventions: Drug: cetuximab + cisplatin + vinorelbine
- Chemotherapy alone (Active Comparator): cisplatin + vinorelbine alone
  Interventions: Drug: cisplatin + vinorelbine

INTERVENTIONS:
Drug: cetuximab + cisplatin + vinorelbine — cetuximab given as an intravenous (i.v.) infusion every week (400mg/m^2 initial dose and 250mg/m^2 subsequent doses) until progressive disease (PD) + cisplatin 80mg/m^2 i.v. infusion on day 1 of each 3-week cycle + vinorelbine 25mg/m^2 i.v. infusion on days 1 and 8 of each 3-week cycle.
  Arms: Cetuximab plus chemotherapy
Drug: cisplatin + vinorelbine — cisplatin 80mg/m^2 i.v. infusion on day 1 of each 3-week cycle + vinorelbine 25mg/m^2 i.v. infusion on days 1 and 8 of each 3-week cycle.
  Arms: Chemotherapy alone

SUMMARY:
The purpose of this trial is to investigate the efficacy of cetuximab in combination with chemotherapy in comparison to chemotherapy alone in patients with advanced non small cell lung cancer who did not received prior chemotherapy. Overall survival will be taken as primary measure of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically confirmed NSCLC, stage IIIb with documented malignant pleural effusion or stage IV
* Immunohistochemical evidence of EGFR expression on tumor tissue
* Presence of at least 1 bi-dimensionally measurable index lesion, whereby index lesions must not lie in an irradiated area

Exclusion Criteria:

* Previous exposure to monoclonal antibodies, signal transduction inhibitors or EGFR-targeting therapy
* Previous chemotherapy for NSCLC
* Documented or symptomatic brain metastasis
* Superior vena cava syndrome contra-indicating hydration
* Previous malignancy in the last 5 years except basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1861 (Actual)
Dates: Start 2004-10; Primary Completion 2007-07 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pirker, Professor, Principal Investigator — Universitätsklinik für Innere Medizin I, Wien
Locations (118):
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Córdoba
- Australia (5):
  - Research Site, Adelaide
  - Research Site, Melbourne
  - Research Site, Randwick
  - Research Site, Sydney
  - Research Site, Wodonga
- Research Site, Vienna, Austria
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Charleroi
  - Research Site, Liège
- Brazil (2):
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Veliko Tarnovo
- Chile (2):
  - Research Site, Antofagasta
  - Research Site, Santiago
- Czechia (4):
  - Research Site, Brno
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Prague
- France (9):
  - Research Site, Brest
  - Research Site, Caen
  - Research Site, Grenoble
  - Research Site, Marseille
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Strasbourg
- Germany (17):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Freiburg im Breisgau
  - Research Site, Gauting
  - Research Site, Göttingen
  - Research Site, Großhansdorf
  - Research Site, Halle-Dölau
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Löwenstein
  - Research Site, Magdeburg
  - Research Site, Mainz
  - Research Site, München
  - Research Site, Stralsund
  - Research Site, Wuppertal
- Research Site, Honh Kong, Hong Kong
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Nyiregyháza
  - Research Site, Székesfehérvár
  - Research Site, Szombathely
  - Research Site, Törökbálint
  - Research Site, Zalegerzeg-Pózva
- Research Site, Dublin, Ireland
- Italy (6):
  - Research Site, Bologna
  - Research Site, Carpi
  - Research Site, Milan
  - Research Site, Rome
  - Research Site, Rozzano-Milano
  - Research Site, Treviglio
- Mexico (2):
  - Research Site, Mexico City
  - Research Site, Monterrey
- Netherlands (3):
  - Research Site, Amsterdam
  - Research Site, Nieuwegeln
  - Research Site, Zwolle
- Poland (6):
  - Research Site, Bydgoszcz
  - Research Site, Olsztyn
  - Research Site, Otwock
  - Research Site, Posnan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Singapore, Singapore
- Slovakia (4):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Nitra-Zobor
  - Research Site, Poprad
- Research Site, Seoul, South Korea
- Spain (11):
  - Research Site, Barakaldo (Bilbao)
  - Research Site, Barcelona
  - Research Site, Donostia / San Sebastian
  - Research Site, Elche Alicante
  - Research Site, Granollers
  - Research Site, Madrid
  - Research Site, Pamplona
  - Research Site, Pontevedra
  - Research Site, Santander
  - Research Site, Terrassa
  - Research Site, Valencia
- Sweden (2):
  - Research Site, Stockholm
  - Research Site, Uppsala
- Switzerland (3):
  - Research Site, Bern
  - Research Site, Thun
  - Research Site, Zurich
- Taiwan (2):
  - Research Site, Taipei, Tao Yuan County
  - Research Site, Taipei
- Research Site, Ankara, Turkey (Türkiye)
- Ukraine (8):
  - Research Site, Dnipropetrovsk
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Poltava
  - Research Site, Sumy
  - Research Site, Ternopil
  - Research Site, Uzhhorod
- United Kingdom (9):
  - Research Site, Aberdeen
  - Research Site, Bristol
  - Research Site, Edinburgh
  - Research Site, Leicester
  - Research Site, London
  - Research Site, Newcastle upon Tyne
  - Research Site, Poole
  - Research Site, Sutton
  - Research Site, Wolverhampton

REFERENCES:
- [Result] Pirker R, Pereira JR, Szczesna A, von Pawel J, Krzakowski M, Ramlau R, Vynnychenko I, Park K, Yu CT, Ganul V, Roh JK, Bajetta E, O'Byrne K, de Marinis F, Eberhardt W, Goddemeier T, Emig M, Gatzemeier U; FLEX Study Team. Cetuximab plus chemotherapy in patients with advanced non-small-cell lung cancer (FLEX): an open-label randomised phase III trial. Lancet. 2009 May 2;373(9674):1525-31. doi: 10.1016/S0140-6736(09)60569-9. PMID 19410716
- [Derived] Pirker R, Pereira JR, Szczesna A, von Pawel J, Krzakowski M, Ramlau R, Vynnychenko I, Park K, Eberhardt WE, de Marinis F, Heeger S, Goddemeier T, O'Byrne KJ, Gatzemeier U. Prognostic factors in patients with advanced non-small cell lung cancer: data from the phase III FLEX study. Lung Cancer. 2012 Aug;77(2):376-82. doi: 10.1016/j.lungcan.2012.03.010. Epub 2012 Apr 11. PMID 22498112
- [Derived] Pirker R, Pereira JR, von Pawel J, Krzakowski M, Ramlau R, Park K, de Marinis F, Eberhardt WE, Paz-Ares L, Storkel S, Schumacher KM, von Heydebreck A, Celik I, O'Byrne KJ. EGFR expression as a predictor of survival for first-line chemotherapy plus cetuximab in patients with advanced non-small-cell lung cancer: analysis of data from the phase 3 FLEX study. Lancet Oncol. 2012 Jan;13(1):33-42. doi: 10.1016/S1470-2045(11)70318-7. Epub 2011 Nov 4. PMID 22056021
- [Derived] O'Byrne KJ, Gatzemeier U, Bondarenko I, Barrios C, Eschbach C, Martens UM, Hotko Y, Kortsik C, Paz-Ares L, Pereira JR, von Pawel J, Ramlau R, Roh JK, Yu CT, Stroh C, Celik I, Schueler A, Pirker R. Molecular biomarkers in non-small-cell lung cancer: a retrospective analysis of data from the phase 3 FLEX study. Lancet Oncol. 2011 Aug;12(8):795-805. doi: 10.1016/S1470-2045(11)70189-9. Epub 2011 Jul 22. PMID 21782507
- [Derived] Gatzemeier U, von Pawel J, Vynnychenko I, Zatloukal P, de Marinis F, Eberhardt WE, Paz-Ares L, Schumacher KM, Goddemeier T, O'Byrne KJ, Pirker R. First-cycle rash and survival in patients with advanced non-small-cell lung cancer receiving cetuximab in combination with first-line chemotherapy: a subgroup analysis of data from the FLEX phase 3 study. Lancet Oncol. 2011 Jan;12(1):30-7. doi: 10.1016/S1470-2045(10)70278-3. Epub 2010 Dec 17. PMID 21169060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/last subject (informed consent): October 2004/January 2006. Clinical data cut-off: 18 July 2007. Last subject completed 16 May 2012. Subjects randomized at 155 centers; Asia/Australia: 21; Europe: 120; South America: 14.
Pre-assignment Details: Enrolled: 1,861 after consent to epidermal growth factor receptor (EGFR) assessment; 603 excluded (mainly non-fulfillment of inclusion or exclusion criteria). 1,258 screened for eligibility after consent for study procedures; 143 excluded (mainly non-fulfillment of inclusion or exclusion criteria). 1,125 subjects randomized.
Groups:
- Cetuximab Plus Chemotherapy: cetuximab given as an intravenous (i.v.) infusion every week (400mg/m^2 initial dose and 250mg/m^2 subsequent doses) until progressive disease (PD) + cisplatin 80mg/m^2 i.v. infusion on day 1 of each 3-week cycle + vinorelbine 25mg/m^2 i.v. infusion on days 1 and 8 of each 3-week cycle.
  Safety population: includes all treated subjects.
- Chemotherapy Alone: cisplatin 80mg/m^2 i.v. infusion on day 1 of each 3-week cycle + vinorelbine 25mg/m^2 i.v. infusion on days 1 and 8 of each 3-week cycle.
  Safety population: includes all treated subjects.
Period: Overall Study
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Started | 557 (Intent To Treat (ITT) Population) | 568 (ITT Population)
Completed | 557 | 568
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone | Total
Number analyzed (Participants) | 557 | 568 | 1125
Age, Continuous [Median (Full Range); unit: years] | 59 [18 to 78] | 60 [20 to 83] | 59 [18 to 83]
Age, Customized [Number; unit: participants]
  <18 years | 0 | 0 | 0
  Between 18 and 65 years | 385 | 389 | 774
  >=65 years | 172 | 179 | 351
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 163 | 335
  Male | 385 | 405 | 790
Region of Enrollment [Number; unit: participants]
  Australia | 20 | 23 | 43
  Hong Kong | 2 | 2 | 4
  Singapore | 5 | 5 | 10
  Korea, Republic of | 28 | 26 | 54
  Taiwan | 21 | 22 | 43
  Austria | 9 | 7 | 16
  Belgium | 3 | 10 | 13
  Bulgaria | 12 | 12 | 24
  Czech Republic | 12 | 17 | 29
  France | 25 | 25 | 50
  Germany | 91 | 88 | 179
  Hungary | 21 | 23 | 44
  Ireland | 3 | 4 | 7
  Netherlands | 10 | 10 | 20
  Poland | 59 | 50 | 109
  Portugal | 3 | 0 | 3
  Russian Federation | 23 | 16 | 39
  Slovakia | 8 | 12 | 20
  Spain | 16 | 13 | 29
  Sweden | 6 | 3 | 9
  Switzerland | 10 | 6 | 16
  Turkey | 1 | 2 | 3
  United Kingdom | 23 | 21 | 44
  Ukraine | 56 | 71 | 127
  Chile | 10 | 16 | 26
  Italy | 18 | 23 | 41
  Argentina | 5 | 2 | 7
  Mexico | 9 | 8 | 17
  Brazil | 48 | 51 | 99

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival Time (OS)
Description: Time from randomization to death. Patients without event are censored at the last date known to be alive or at the clinical cut-off date, whatever is earlier.
Time Frame: Time from randomisation to death or last day known to be alive, reported between day of first patient randomised, Oct 2004, until cut-off date 18 Jul 2007
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 557 | 568
months | 11.3 [9.4 to 12.4] | 10.1 [9.1 to 10.9]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; Primary efficacy analysis: To test equality of OS time between treatment groups, applying the two-sided stratified log-rank test (Stage IIIb vs IV, ECOG 0/1 vs 2) (α=5%); Test type: Superiority or Other; p = 0.0441, Stratified Log Rank

2. Secondary Outcome: Progression-free Survival Time
Description: Duration from randomization until radiological progression (based on modified World Health Organisation (WHO) criteria) or death due to any cause.
  Only deaths within 60 days of last tumor assessment are considered. Patients without event are censored on the date of last tumor assessment.
Time Frame: Time from randomization to disease progression, death or last tumor assessment, reported between day of first patient randomised, Oct 2004, until cut-off date 18 Jul 2007
Population: ITT
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 557 | 568
months | 4.8 [4.2 to 5.3] | 4.8 [4.4 to 5.4]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; To test equality of progression free survival time between treatment groups, applying the two-sided stratified log-rank test (α=5%); Test type: Superiority or Other; p = 0.3869, Stratified Log Rank

3. Secondary Outcome: Best Overall Response Rate
Description: The best overall response rate is defined as the proportion of subjects having achieved confirmed Complete Response + Partial Response as the best overall response according to radiological assessments (based on modified WHO criteria).
Time Frame: Evaluations were performed every 6 weeks until progression, reported between day of first patient randomised, Oct 2004, until cut-off date 18 Jul 2007
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 557 | 568
percentage of participants | 36.4 [32.4 to 40.6] | 29.2 [25.5 to 33.2]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; The best overall response rate was compared in the Cochran-Mantel-Haenszel test (two-sided with α=5%); Test type: Superiority or Other; p = 0.0101, Cochran-Mantel-Haenszel

4. Secondary Outcome: Disease Control Rate
Description: The disease control rate is defined as the proportion of subjects having achieved confirmed Complete Response + Partial Response + Stable Disease as best overall response according to radiological assessments (based on modified WHO criteria).
Time Frame: as for outcome 3
Population: ITT
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 557 | 568
percentage of participants | 72.5 [68.6 to 76.2] | 71.5 [67.6 to 75.2]
Statistical Analysis 1: Comparison: Cetuximab Plus Chemotherapy vs Chemotherapy Alone; The disease control rate was compared in the Cochran-Mantel-Haenszel test (two-sided with α=5%); Test type: Superiority or Other; p = 0.6801, Cochran-Mantel-Haenszel

5. Secondary Outcome: Quality of Life (QOL) Assessment European Organisation for the Research and Treatment of Cancer (EORTC) QLQ-C30 Global Health Status
Description: Mean global health status scores (EORTC QLQ-C30) against time for each treatment group. Scores were derived from mutually exclusive sets of items, with scale scores ranging from 0 to 100 after a linear transformation. Higher scores indicate a better QoL.
Time Frame: at baseline, at cycle 3, at month 6, reported between day of first patient randomised, Oct 2004, until cut-off date 18 Jul 2007
Population: 670 subjects completed (348 in the cetuximab + chemotherapy arm and 322 in the chemotherapy alone arm) at least 1 evaluable QLQ-C30 questionnaire and were included in the Evaluable population. Numbers at each timepoint were (Cetuximab + chemotherapy/Chemotherapy alone, respectively): baseline 278/274; cycle 3 184/153; 6 month 102/96
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 348 | 322
scores on a scale
  At baseline | 45.72 (2.164) | 46.36 (2.138)
  At cycle 3 | 48.33 (2.325) | 51.55 (2.464)
  At month 6 | 54.71 (2.729) | 52.92 (2.787)

6. Secondary Outcome: Quality of Life Assessment (EORTC QLQ-C30) Social Functioning
Description: Mean social functioning scores (EORTC QLQ-C30) against time for each treatment group. Scores were derived from mutually exclusive sets of items, with scale scores ranging from 0 to 100 after a linear transformation. Higher scores indicate a higher level of functioning.
Time Frame: as for outcome 5
Population: 670 subjects completed (348 in the cetuximab + chemotherapy arm and 322 in the chemotherapy alone arm) at least 1 evaluable QLQ-C30 questionnaire and were included in the Evaluable population. Numbers at each timepoint were (Cetuximab + chemotherapy/Chemotherapy alone, respectively): baseline 280/275; cycle 3 185/153; 6 month 101/97
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 348 | 322
scores on a scale
  At baseline | 66.17 (2.836) | 64.73 (2.825)
  At cycle 3 | 58.05 (2.995) | 67.13 (3.138)
  At month 6 | 67.36 (3.449) | 66.47 (3.515)

7. Secondary Outcome: A Population Pharmacokinetic (PK) Analysis for Cetuximab in Non-Small Cell Lung Cancer (NSCLC) - Serum Cetuximab Concentrations
Description: Population PK analysis was conducted using non-linear mixed effects modeling (NONMEM) software, integrating the PK data from this study and the Phase II study EMR 62 202-011.
Time Frame: Week 1, Day 1: baseline and end of infusion; Week 7, Day 43: within 12 h after cetuximab administration.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Cetuximab Concentration at End of Infusion Week 1 | Cetuximab Concentration Before Infusion Week 7
Number analyzed (Participants) | 454 | 298
ug/mL | 223.1 (64.6) | 51.5 (33.1)

8. Secondary Outcome: Safety - Number of Patients Experiencing Any Adverse Event
Description: Please refer to Adverse Events section for further details
Time Frame: time from first dose up to 30 after last dose of study treatment, reported between day of first patient randomised, Oct 2004, until cut-off date 18 Jul 2007
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Number analyzed (Participants) | 548 | 562
participants | 545 | 549

ADVERSE EVENTS:
Time Frame: Time from first dose up to 30 days after the last dose of study treatment.
Description: Treatment-emergent adverse events were defined as those with onset occurring at or after the first dosing day of study medication and up to 30 days after the last administration of any study drug or the clinical cut-off date.
Arm/Group | Cetuximab Plus Chemotherapy | Chemotherapy Alone
Serious Adverse Events (participants affected / at risk) | 325/548 | 244/562
Other Adverse Events (participants affected / at risk) | 532/548 | 537/562
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Chemotherapy (N=548) | Chemotherapy Alone (N=562)
Anaemia (Blood and lymphatic system disorders) | 11 | 12
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 4 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 96 | 67
Granulocytopenia (Blood and lymphatic system disorders) | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 15 | 8
Neutropenia (Blood and lymphatic system disorders) | 47 | 33
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 4 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 4
Cardiac arrest (Cardiac disorders) | 0 | 2
Cardiac failure (Cardiac disorders) | 1 | 2
Cardiac failure acute (Cardiac disorders) | 2 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 3 | 3
Left ventricular failure (Cardiac disorders) | 2 | 0
Microvascular angina (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 2 | 2
Right ventricular failure (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 1
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Tracheo-oesophageal fistula (Congenital, familial and genetic disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 8
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 8 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Haematemesis (Gastrointestinal disorders) | 2 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 5
Odynophagia (Gastrointestinal disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 16 | 14
Asthenia (General disorders) | 4 | 2
Chest discomfort (General disorders) | 0 | 2
Chest pain (General disorders) | 7 | 6
Death (General disorders) | 2 | 0
Drug interaction (General disorders) | 1 | 0
Fatigue (General disorders) | 5 | 2
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 22 | 4
Injection site reaction (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 2 | 1
Multi-organ failure (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 16 | 6
Sudden death (General disorders) | 2 | 0
Hepatic pain (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 0
Anaphylactic reaction (Immune system disorders) | 3 | 0
Anaphylactic shock (Immune system disorders) | 2 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 5 | 1
Serum sickness (Immune system disorders) | 1 | 0
Anal abscess (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 2 | 2
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 1
Catheter related infection (Infections and infestations) | 3 | 0
Cellulitis (Infections and infestations) | 4 | 0
Central line infection (Infections and infestations) | 1 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Dengue fever (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 3 | 1
Laryngitis (Infections and infestations) | 1 | 0
Laryngotracheo bronchitis (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 4 | 2
Lung abscess (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 9 | 5
Neutropenic sepsis (Infections and infestations) | 9 | 5
Parotitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pharyngotonsillitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 19 | 13
Pneumonia necrotising (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Pyothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 2
Sepsis (Infections and infestations) | 9 | 3
Septic shock (Infections and infestations) | 6 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Aspiration bronchial (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 5 | 4
Blood glucose abnormal (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood urea increased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 2 | 0
Karnofsky scale worsened (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Pulmonary arterial pressure increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 2 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 12 | 9
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypercreatininaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Testis cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Cerebral infarction (Nervous system disorders) | 0 | 2
Cerebral ischaemia (Nervous system disorders) | 3 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 5
Cognitive disorder (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 3 | 0
Coordination abnormal (Nervous system disorders) | 1 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 0 | 1
Embolic cerebral infarction (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Horner's syndrome (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 2
Paraplegia (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 2 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 2
Syncope vasovagal (Nervous system disorders) | 1 | 1
Transverse sinus thrombosis (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 5 | 4
Depression (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 1
Mental disorder (Psychiatric disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 6 | 6
Renal failure acute (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 13
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 20 | 13
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 14 | 9
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 0 | 2
Arterial thrombosis (Vascular disorders) | 1 | 0
Axillary vein thrombosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 9 | 3
Embolism (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 5 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Pelvic venous thrombosis (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 0 | 2
Shock (Vascular disorders) | 1 | 0
Superior vena caval occlusion (Vascular disorders) | 1 | 2
Thrombosis (Vascular disorders) | 2 | 2
Varicose vein (Vascular disorders) | 0 | 1
Vascular fragility (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 1
Visceral arterial ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab Plus Chemotherapy (N=548) | Chemotherapy Alone (N=562)
Neutropenia (Blood and lymphatic system disorders) | 302 | 324
Anaemia (Blood and lymphatic system disorders) | 226 | 264
Leukopenia (Blood and lymphatic system disorders) | 176 | 155
Febrile neutropenia (Blood and lymphatic system disorders) | 36 | 32
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 30
Tinnitus (Ear and labyrinth disorders) | 49 | 55
Conjunctivitis (Eye disorders) | 33 | 6
Nausea (Gastrointestinal disorders) | 291 | 303
Vomiting (Gastrointestinal disorders) | 214 | 225
Constipation (Gastrointestinal disorders) | 204 | 189
Diarrhoea (Gastrointestinal disorders) | 126 | 103
Stomatitis (Gastrointestinal disorders) | 85 | 27
Abdominal pain (Gastrointestinal disorders) | 72 | 72
Dyspepsia (Gastrointestinal disorders) | 68 | 55
Abdominal pain upper (Gastrointestinal disorders) | 45 | 37
Dysphagia (Gastrointestinal disorders) | 31 | 7
Fatigue (General disorders) | 202 | 181
Pyrexia (General disorders) | 112 | 80
Asthenia (General disorders) | 90 | 96
Chest pain (General disorders) | 70 | 70
Mucosal inflammation (General disorders) | 56 | 23
Chills (General disorders) | 35 | 19
Injection site reaction (General disorders) | 33 | 29
Oedema peripheral (General disorders) | 29 | 39
Paronychia (Infections and infestations) | 46 | 0
Nasopharyngitis (Infections and infestations) | 37 | 16
Weight decreased (Investigations) | 75 | 50
Blood creatinine increased (Investigations) | 47 | 49
White blood cell count decreased (Investigations) | 36 | 26
Anorexia (Metabolism and nutrition disorders) | 208 | 202
Hypokalaemia (Metabolism and nutrition disorders) | 75 | 49
Hypomagnesaemia (Metabolism and nutrition disorders) | 54 | 27
Hypocalcaemia (Metabolism and nutrition disorders) | 31 | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 53 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 39 | 44
Myalgia (Musculoskeletal and connective tissue disorders) | 39 | 37
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 22
Bone pain (Musculoskeletal and connective tissue disorders) | 29 | 28
Dizziness (Nervous system disorders) | 82 | 57
Headache (Nervous system disorders) | 79 | 60
Peripheral sensory neuropathy (Nervous system disorders) | 49 | 46
Paraesthesia (Nervous system disorders) | 40 | 27
Dysgeusia (Nervous system disorders) | 31 | 33
Insomnia (Psychiatric disorders) | 58 | 49
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 101 | 95
Cough (Respiratory, thoracic and mediastinal disorders) | 97 | 80
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 45 | 24
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 33 | 14
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 31 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 30 | 15
Rash (Skin and subcutaneous tissue disorders) | 249 | 17
Alopecia (Skin and subcutaneous tissue disorders) | 107 | 107
Dry skin (Skin and subcutaneous tissue disorders) | 76 | 9
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 75 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 64 | 13
Acne (Skin and subcutaneous tissue disorders) | 38 | 2
Skin fissures (Skin and subcutaneous tissue disorders) | 30 | 0
Phlebitis (Vascular disorders) | 48 | 44
Hypertension (Vascular disorders) | 40 | 27
Hypotension (Vascular disorders) | 39 | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other